CLINICAL TRIAL: NCT04165772
Title: A Phase II Study of Induction PD-1 Blockade in Subjects With Locally Advanced Mismatch Repair Deficient Solid Tumors
Brief Title: Study of Induction PD-1 Blockade in Subjects With Locally Advanced Mismatch Repair Deficient Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-288
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Rectal Adenocarcinoma; Clinical Stage: Stage II (T3-4, N-); Stage III (Any T, N+); Solid Tumor; Solid Tumor, Adult
Keywords: PD1 blockade; TSR-042; Radiation; Capecitabine; 5-FU; 19-288; Solid tumor; Dostarlimab
MeSH Terms: conditions — Rectal Neoplasms | interventions — dostarlimab; Capecitabine; Fluorouracil; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: This is a Phase II study investigating the efficacy of PD1 blockade with TSR-042 in patients with locally advanced MMRd or MSI rectal adenocarcinoma.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Patients with clinical Stage II or Stage III MRI-staged, MSI-H or dMMR, solid tumors will receive up to 6 months (9, 21-day cycles) of PD-1 blockade followed by radiological and surgical restaging of the tumor. If subject exhibits complete clinical response, non-operative management will be followed. If a complete clinical response is not reached after 6 months of PD-1 blockade, the participant will proceed with standard chemoradiation. After completing chemoradiation participant will be assessed for response if complete CR is not obtained then the participant will proceed with disease specific surgical resection or standard of care therapy.
  Interventions: Drug: TSR-042 or Dostarlimab; Drug: capecitabine or 5-FU; Radiation: Intensity Modulated Radiation Therapy (IMRT)
- Cohort 2 (Other): The plan is to enroll six patients with MSI, regardless of their primary cancer diagnosis. This cohort will serve to generate hypothesis and initial data to plan a larger study. All analyses from this cohort will be exploratory
  Interventions: Drug: TSR-042 or Dostarlimab

INTERVENTIONS:
Drug: TSR-042 or Dostarlimab — Patients will be given TSR-042/Dostarlimab at a dose of 500mg IV, over 30 minutes Q 3 weeks.
  Other Names: Dostarlimab
Drug: capecitabine or 5-FU — Capecitabine 825mg/m2 BID concurrently with radiation per standard radiation guidelines. If patient is unable to tolerate oral medication, infusional 5-FU is an acceptable alternative.
  Arms: Cohort 1
Radiation: Intensity Modulated Radiation Therapy (IMRT) — The radiation dose is 5400 cGy to the tumor and surrounding nodes 4700 cGy to the pelvis, with an integrated boost to the primary tumor and involved nodes of receiving 5400cGy in 27fx.
  Arms: Cohort 1

SUMMARY:
The purpose of this study is to find out whether the study drug, TSR-042, followed by standard chemoradiotherapy (the chemotherapy drug capecitabine + radiation therapy) and standard surgery is an effective treatment for advanced dMMR solid tumors. The study will also look at the safety of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for the trial.
* Be ≥18 years of age on the date of signing informed consent.
* ECOG performance status of 0 or 1.
* Histologically confirmed locally advanced solid tumor
* Solid tumors that in standard practice would be treated with neoadjuvant therapy
* No evidence of distant metastases.

  * Radiologically measurable or clinically evaluable disease
* Tumor specimen that demonstrates mismatch repair deficiency by Immunohistochemistry or microsatellite instability as demonstrated by NGS or PCR.
* Negative pregnancy test done 72 hours prior to beginning treatment, for women of childbearing potential only. Subjects of childbearing potential must be willing to use an adequate method of contraception. Appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives, or double barrier method (diaphragm plus condom). Contraception, for the course of the study starting with the first dose of study medication through 150 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Nonchildbearing potential is defined as follows (by other than medical reasons):

* ≥45 years of age and has not had menses for >1 year
* Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
* Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study.

  * Participant receiving corticosteroids may continue if their dose is stable for least 4 weeks prior to initiating protocol therapy.
  * Has QTcF ≤ 450 msec, or ≤ 480 msec for participants with bundle branch block.
  * Demonstrate adequate organ function as defined below within 14 days of Cycle 1, Day 1, all screening labs should be performed within 14 days of treatment initiation.
  * Hematological
* Absolute neutrophil count (ANC) ≥1,500 /mcL
* Platelets ≥100,000 / mcL
* Hemoglobin >9 g/dL or ≥5.6 mmol/L

  * Renal
* Serum creatinine OR Measured or calculated(a) creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 × institutional ULN

  * Hepatic
* Serum total bilirubin ≤ 1.5 × ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN

  * Coagulation
* International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended (a) Creatinine clearance should be calculated per institutional standard.

Exclusion Criteria:

* Presence of metastatic or recurrent disease
* Prior radiation therapy, chemotherapy, or surgery for tumor
* For patients with colorectal primary -Tumor is causing symptomatic bowel obstruction (patients who have a temporary diverting ostomy are eligible).
* Cohort 1 Only: Other invasive malignancy ≤ 5 years prior to registration. Exceptions are non-melanoma skin cancer that has undergone potentially curative therapy and in situ cervical carcinoma.
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of non- physiologic dose immunosuppressive therapy within 7 days prior to first dose of trial treatment.
* Active autoimmune disease requiring systemic treatment within the past 2 years or documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents at non-physiologic doses.
* Active infection requiring systemic therapy.
* Cohort 1 Only: Received prior therapy with an antibody or drug specifically targeting T- cell co-stimulation or checkpoint pathways.
* Experienced ≥ Grade 3 immune-related AE with prior immunotherapy, except for non-clinically significant lab abnormalities.
* Other Anticancer or Experimental Therapy. No other experimental therapies (including chemotherapy, radiation, hormonal treatment, antibody therapy, immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, matrix metalloprotease inhibitors, thalidomide, anti-VEGF/Flk-1 monoclonal antibody or other experimental drugs) of any kind are permitted while the patient is receiving study treatment.
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Women who are pregnant or breastfeeding, or men expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening visit through 150 days after the last dose of study medication.
* Concurrent medical or psychiatric condition or disease which, in the investigator's judgement, would make them inappropriate candidates for entry into the study. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, chronic obstructive pulmonary disease, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
* Received a live vaccine within 30 days of planned start of study medication.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment.
* History of interstitial lung disease.
* Known hypersensitivity to TSR-042 components or excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) or complete clinical response (cCR) at 12 months | 12 months
  To determine the pathologic complete response rate (pCR) or complete clinical response (cCR) rate at 12 months, after PD-1 blockade and with or without chemoradiation in subjects with mismatch repair deficient locally advanced adenocarcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cercek, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Hartford Healthcare (Data Collection), Hartford, Connecticut
  - Baptist Alliance MCI (Data Collection Only), Miami, Florida
  - Memorial Sloan Kettering Basking Ridge - Limited Protocol Activities, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth - Limited Protocol Activities, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen - Limited Protocol Activities, Montvale, New Jersey
  - Memorial Sloan Kettering Commack - Limited Protocol Activities, Commack, New York
  - Memorial Sloan Kettering Westchester - Limited Protocol Activities, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau - Limited Protocol Activities, Uniondale, New York
  - Lehigh Valley Health Network (Data Collection Only), Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Cercek A, Foote MB, Rousseau B, Smith JJ, Shia J, Sinopoli J, Weiss J, Lumish M, Temple L, Patel M, Wilde C, Saltz LB, Argiles G, Stadler Z, Artz O, Maron S, Ku G, Gu P, Janjigian YY, Molena D, Iyer G, Coleman J, Abida W, Cohen S, Soares K, Schattner M, Strong VE, Yaeger R, Paty P, Shcherba M, Sugarman R, Romesser PB, Zervoudakis A, Desai A, Segal NH, El Dika I, Widmar M, Wei I, Pappou E, Fumo G, Aparo S, Gonen M, Gollub M, Jayaprakasam VS, Kim TH, Garcia Aguilar J, Weiser M, Diaz LA Jr. Nonoperative Management of Mismatch Repair-Deficient Tumors. N Engl J Med. 2025 Jun 19;392(23):2297-2308. doi: 10.1056/NEJMoa2404512. Epub 2025 Apr 27. PMID 40293177
- [Derived] Saude-Conde R, Nguyen D, Hendlisz A. Immunotherapies in non-metastatic gastrointestinal cancers. Curr Opin Oncol. 2023 Jul 1;35(4):334-346. doi: 10.1097/CCO.0000000000000956. Epub 2023 May 9. PMID 37222204
- [Derived] Costa B, Vale N. Dostarlimab: A Review. Biomolecules. 2022 Jul 26;12(8):1031. doi: 10.3390/biom12081031. PMID 35892341
- [Derived] Cercek A, Lumish M, Sinopoli J, Weiss J, Shia J, Lamendola-Essel M, El Dika IH, Segal N, Shcherba M, Sugarman R, Stadler Z, Yaeger R, Smith JJ, Rousseau B, Argiles G, Patel M, Desai A, Saltz LB, Widmar M, Iyer K, Zhang J, Gianino N, Crane C, Romesser PB, Pappou EP, Paty P, Garcia-Aguilar J, Gonen M, Gollub M, Weiser MR, Schalper KA, Diaz LA Jr. PD-1 Blockade in Mismatch Repair-Deficient, Locally Advanced Rectal Cancer. N Engl J Med. 2022 Jun 23;386(25):2363-2376. doi: 10.1056/NEJMoa2201445. Epub 2022 Jun 5. PMID 35660797
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm